CLINICAL TRIAL: NCT01203267
Title: Phase 2 Study of Weekly Paclitaxel Plus Carboplatin in Preoperative Treatment of Breast Cancer Patients
Brief Title: Weekly Paclitaxel Plus Carboplatin in Preoperative Treatment of Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Fudan University (Other); Ruijin Hospital (Other)
Responsible Party: Kunwei Shen/Shanghai Jiao Tong University, Shanghai Jiao Tong University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DXK200801
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2007-11

CONDITIONS: Breast Cancer
Keywords: Breast Neoplasms; Neoadjuvant; Chemotherapy; Paclitaxel; Carboplatin; Pathological Complete Remission
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response | interventions — CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- paclitaxel plus carboplatin (PCb) Arm (Experimental): 4 cycles of neoadjuvant paclitaxel plus carboplatin
  Interventions: Drug: Paclitaxel, Carboplatin

INTERVENTIONS:
Drug: Paclitaxel, Carboplatin — Paclitaxel 80 mg/m2, carboplatin AUC of 2 mg/min/ml, given on days 1, 8 and 15 of a 28-day cycle.

SUMMARY:
The purpose of this study is to evaluate the pathological complete response (pCR) rate in breast cancer patients treated with weekly paclitaxel plus carboplatin preoperative regimen.

DETAILED DESCRIPTION:
Breast cancer is the leading cause of cancer in women in China. Preoperative chemotherapy for treatment of locally advanced breast cancer has become a standard therapy. Results from neoadjuvant trials have shown that pathological complete response (pCR) is an independent predictor of outcome. Paclitaxel was introduced into clinical practice in the early 1990s and has demonstrated good activity in the adjuvant and metastatic settings. Platinum complexes, like cisplatin and carboplatin, are active in a wide range of solid tumors. Paclitaxel combined with carboplatin has shown great activity in ovarian and nonsmall- cell lung cancer treatment. In addition, the overall response rate of paclitaxel plus carboplatin was between 53% and 62% in the first-line treatment of metastatic breast cancer. This study will evaluate the pCR rate of weekly paclitaxel plus carboplatin as preoperative treatment for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years and < 70 years
* Karnofsky performance status (KPS) ≥ 70
* At least one measurable disease according to the RECIST. histologically confirmed invasive breast cancer (excluding inflammatory breast cancer), large operable (T≥3 cm and N0-1) or locally advanced breast cancer (T3-4N0-3 or T0-4N2-3)
* Biopsy specimens are available for ER, PgR and Her2 analysis
* Adequate bone marrow function: Neutrophil ≥ 1.5*109/L; Hb ≥ 100g/L; PLT ≥ 100*109/L
* An estimated life expectancy of at least 12 months
* Willing to take biopsy before neoadjuvant chemotherapy and patients must be accessible for treatment and follow-up
* Women with potential child-bearing must have a negative pregnancy test (urine or serum) within 7 days of drug administration and agree to use an acceptable method of birth control to avoid pregnancy for the duration of the study
* Written informed consent according to the GCP

Exclusion Criteria:

* Prior systemic or loco-regional treatment of breast cancer, including chemotherapy
* Metastatic breast cancer
* With a history of malignant tumor except uterine cervix cancer in situ or skin basal cell carcinoma
* Patients with medical conditions that indicate intolerant to neoadjuvant therapy and related treatment, including uncontrolled pulmonary disease, diabetes mellitis, severe infection, active peptic ulcer, coagulation disorder, connective tissue disease or myelo-suppressive disease
* inadequate liver function (bilirubin > 1.0 times upper normal limit [UNL] and ALT and/or AST> 1.5 UNL associated with alkaline phosphatase > 2.5 UNL; inadequate renal function (creatinine > 1.0 times UNL and in case of limit value, Creatinine clearance < 60 ml/min)
* Contraindication for using dexamethasone
* History of congestive heart failure, uncontrolled or symptomatic angina pectoris, arrhythmia or myocardial infarction; poorly controlled hypertension (systolic BP > 180 mmHg or diastolic BP > 100 mmHg)
* Has peripheral neuropathy ≥ grade 1
* Patient is pregnant or breast feeding
* Known severe hypersensitivity to any drugs in this study
* Treatment with any investigational drugs within 30 days before the beginning of study treatment

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
pathological complete remission (pCR) rate | after 4 cycles of preoperative treatment

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 4 months during neoadjuvant therapy
  From the first dose of neoadjuvant chemotherapy to definitive surgery or disease progression
clinical response rate | after 4 cycles of preoperative therapy
Predictive markers of weekly paclitaxel plus carboplatin | after 4 cycles of preoperative treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kunwei Shen, Dr, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Yang L, Li LD, Chen YD, Parkin DM. [Time trends, estimates and projects for breast cancer incidence and mortality in China]. Zhonghua Zhong Liu Za Zhi. 2006 Jun;28(6):438-40. Chinese. PMID 17152490
- [Background] Rouzier R, Perou CM, Symmans WF, Ibrahim N, Cristofanilli M, Anderson K, Hess KR, Stec J, Ayers M, Wagner P, Morandi P, Fan C, Rabiul I, Ross JS, Hortobagyi GN, Pusztai L. Breast cancer molecular subtypes respond differently to preoperative chemotherapy. Clin Cancer Res. 2005 Aug 15;11(16):5678-85. doi: 10.1158/1078-0432.CCR-04-2421. PMID 16115903
- [Background] Frasci G, Comella P, Rinaldo M, Iodice G, Di Bonito M, D'Aiuto M, Petrillo A, Lastoria S, Siani C, Comella G, D'Aiuto G. Preoperative weekly cisplatin-epirubicin-paclitaxel with G-CSF support in triple-negative large operable breast cancer. Ann Oncol. 2009 Jul;20(7):1185-92. doi: 10.1093/annonc/mdn748. Epub 2009 Feb 13. PMID 19218307
- [Result] Chen XS, Nie XQ, Chen CM, Wu JY, Wu J, Lu JS, Shao ZM, Shen ZZ, Shen KW. Weekly paclitaxel plus carboplatin is an effective nonanthracycline-containing regimen as neoadjuvant chemotherapy for breast cancer. Ann Oncol. 2010 May;21(5):961-7. doi: 10.1093/annonc/mdq041. Epub 2010 Mar 8. PMID 20211870